CLINICAL TRIAL: NCT06232317
Title: Feasibility and Acceptability of ReCognitionVR-based Cognitive Stimulation in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hina Faisal, Assistant Professor of Clinical Surgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00037724; R03AG078857 (NIH)
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Surgery; Delirium; Delirium, Post-Operative
Keywords: abdominal surgery; virtual reality
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Software (Experimental): Participants in this arm will receive cognitive exercises using ReCognitionVR virtual reality software
  Interventions: Other: Virtual Reality Software
- Traditional Orientation Methods (Active Comparator): Participants in this arm will receive cognitive exercises using traditional (standard-of-care) orientation methods,
  Interventions: Other: Traditional Orientation Methods

INTERVENTIONS:
Other: Virtual Reality Software — The ReCognitionVR virtual reality software is delivered via an Oculus Quest 2 device. This three-dimensional simulated software was designed to improve attention and executive functions.
  Other Names: ReCognitionVR
  Arms: Virtual Reality Software
Other: Traditional Orientation Methods — Standard-of-care methods to orient patients after surgery
  Arms: Traditional Orientation Methods

SUMMARY:
This study aims to assess the feasibility, acceptability, and safety of using ReCognitionVR virtual reality-based software in older surgical patients. Results from this study will be used to inform the design of a future study in critically ill hospitalized patients at risk for delirium.

DETAILED DESCRIPTION:
Virtual reality (VR) imitates reality by creating an artificial 3-dimensional (3D) environment using computing technology or software. A virtual environment (VE) is created using this software with a headset, which cognitively stimulates the user's brain to think they are in an artificial world. Creating a VE allows flexibility and measurement of different types of stimuli while recording the various responses provided by users in the controlled VE. VR strengthens the brain's ability to focus, learn, and retain experience. VR for attention deficit disorders has been reported to have promising results. We followed in similar footsteps and designed and developed a novel, 3D simulated software platform prototype called ReCognition VR to provide VR-based cognitive exercises.

A feasibility clinical trial conducted by our group tested the ReCognitionVR cognitive interventions on older and young healthy volunteers (NCT05583903). The results of this study showed that ReCognitionVR-based cognitive exercises were feasible, acceptable, and tolerable by older healthy subjects. In stage 2 of our research study, we want to evaluate the safety, feasibility, acceptability, and tolerability of VR-based cognitive exercises in 60-year-old or older patients following abdominal surgery admitted to the surgical floor at Houston Methodist Hospital (HMH). Our premise is that VR-based cognitive stimulation software will allow the controlled delivery of structured cognitive exercises focusing on orientation, attention, memory, and executive functions. The system will allow customized frequency and duration of cognitive exercises based on the users' difficulty level in a delightfully relaxed environment with beach wave sounds.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 years of age
* Scheduled to undergo the following abdominal surgeries (open or laparoscopic or robotic assisted): small bowel and large bowel surgery; cholecystectomy; Whipple procedure; pancreatectomy; splenectomy.
* Richmond Agitation-Sedation Scale (RASS) Score 0

Exclusion Criteria:

* Subjects with baseline cognitive impairment
* Person with active psychiatric disorders and being treated with medications, especially schizophrenia
* Person who is deaf or blind
* Person with an underlying cognitive disorder or associated phobias (e.g., claustrophobia)
* Person participating in other clinical trials involving drugs, biologics, devices, or behavioral interventions
* Active seizure disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hina Faisal, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality Software | Traditional Orientation Methods | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (5) | 69 (5) | 67 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 9 | 13 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.21 (4.32) | 26.38 (6.08) | 27.30 (5.27)
Active smoker [Count of Participants; unit: Participants]
  Yes | 5 | 6 | 11
  No | 10 | 9 | 19
History of hypertension [Count of Participants; unit: Participants] | 10 | 10 | 20
History of diabetes [Count of Participants; unit: Participants] | 3 | 4 | 7
History of hypercholesterolemia [Count of Participants; unit: Participants] | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Treatment-emergent Adverse Events (TEAE)
Description: Percentage of participants who experience a treatment-emergent adverse event (TEAE) in the virtual reality software (experimental) arm compared to the Traditional Orientation Methods (control) arm.
Time Frame: Within 1 month of enrolling in the study
Measure: Number; unit: percent
Groups:
- Traditional Orientation Methods (Control): Patients randomized to the traditional orientation method, were visited by a nurse at the start of each nursing shift. The nurse asked them questions to check their memory and attention. Examples of questions include asking the patient for their name, the date, where they were, and what just happened to them. This will be repeated during every nurse shift change and is the usual care they would receive, even if they were not in the study.
Arm/Group | Virtual Reality Software | Traditional Orientation Methods (Control)
Number analyzed (Participants) | 15 | 15
percent | 0 | 0

2. Secondary Outcome: Change From Baseline in Pulse Oximetry Oxygen Saturation After 10 Minutes
Description: Pulse oximetry oxygen saturation measured using a vital sign monitor at baseline (immediately prior to VR software use and 10 minutes after VR software use. Change = 10-minute oxygen saturation - baseline oxygen saturation
Time Frame: Baseline and 10 minutes
Population: This analysis was only performed for the experimental arm because participants in the active comparator arm (traditional orientation methods) were not exposed to the virtual reality software
Measure: Mean (Standard Deviation); unit: percent oxygen saturation
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
percent oxygen saturation | -1 (2)

3. Secondary Outcome: Change From Baseline in Respiratory Rate After 10 Minutes
Description: Respiratory rate at baseline (immediately prior to virtual reality software use and 10 minutes after use. Change = 10-minute respiratory rate - baseline respiratory rate
Time Frame: Baseline and 10 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
breaths per minute | 0 (0)

4. Secondary Outcome: Change From Baseline in Systolic Blood Pressure After 10 Minutes
Description: Systolic blood pressure measured using a vital sign monitor at baseline (immediately prior to virtual reality software use) and 10 minutes after software use. Change = 10-minute systolic blood pressure - baseline systolic blood pressure
Time Frame: Baseline and 10 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
mm Hg | 3.93 (11.32)

5. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure After 10 Minutes
Description: Diastolic blood pressure measured using a vital sign monitor at baseline (immediately prior to virtual reality software use) and 10 minutes after software use. Change = 10-minute diastolic blood pressure - baseline diastolic blood pressure
Time Frame: Baseline and 10 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
mm Hg | 2.33 (4.55)

6. Secondary Outcome: Change From Baseline in Pulse Oximetry Oxygen Saturation After Completion
Description: Pulse oximetry oxygen saturation measured using a vital sign monitor at baseline (immediately prior to virtual reality software use) and after completion of software use. Change = completion oxygen saturation - baseline oxygen saturation
Time Frame: Baseline and completion of the intervention, up to 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent oxygen saturation
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
percent oxygen saturation | -0.47 (1.85)

7. Secondary Outcome: Change From Baseline in Respiratory Rate After Completion
Description: Respiratory rate at baseline (immediately prior to virtual reality software use) and after software use. Change = completion respiratory rate - baseline respiratory rate
Time Frame: Baseline and completion of the intervention, up to 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
breaths per minute | 0 (0)

8. Secondary Outcome: Change From Baseline in Systolic Blood Pressure After Completion
Description: Systolic blood pressure measured using a vital sign monitor at baseline (immediately prior to virtual reality software use) and after completion of software use. Change = completion systolic blood pressure - baseline systolic blood pressure
Time Frame: Baseline and completion of the intervention, up to 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
mm Hg | -6.27 (13.49)

9. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure After Completion
Description: Diastolic blood pressure measured using a vital sign monitor at baseline (immediately prior to virtual reality software use) and after software use. Change = completion diastolic blood pressure - baseline diastolic blood pressure
Time Frame: Baseline and completion of the intervention, up to 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
mm Hg | -1.40 (6.79)

10. Secondary Outcome: Positive Confusion Assessment Method and/or 4 A's Test
Description: The proportion of patients who have a positive Confusion Assessment Method (CAM) or 4 A's Test for delirium
Time Frame: Baseline to discharge from hospital, up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

11. Secondary Outcome: Change in Visual Analog Scale (VAS) Pain Score
Description: Change in VAS pain score using numeric pain rating scale, where 0 is minimum (no pain) and 10 is maximum (highest pain), from start of intervention to end of intervention (experimental arm) or enrollment to 24 hours post-enrollment (control arm)
Time Frame: Enrollment in study to 24 hours after study enrollment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
Number analyzed (Participants) | 15 | 15
score on a scale | 0 [-1 to 0] | 0 [-2 to 1]
Statistical Analysis 1: Comparison: Virtual Reality Software vs Traditional Orientation Methods; Test type: Superiority; p = 0.61, Kruskal-Wallis

12. Secondary Outcome: Change in Virtual Analog Scale (VAS) Pain Score Value Beginning to Mid-intervention
Description: Change in VAS pain score using numeric pain rating scale, where 0 is minimum (no pain) and 10 is maximum (highest pain), from pre-virtual reality use to 10 minutes after beginning use (experimental arm) or enrollment to 8-16 hours post-enrollment (control arm)
Time Frame: Virtual Reality Software arm: 10 minutes after beginning use; Traditional Orientation Methods arm: 8-16 hours after enrollment (one measure, window allowed for completing the measure)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
Number analyzed (Participants) | 15 | 15
score on a scale | 0 [-1 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Virtual Reality Software vs Traditional Orientation Methods; Test type: Superiority; p = 0.014, Kruskal-Wallis

13. Other Pre Specified Outcome: Percentage of Participants Using Virtual Reality Software at 20 Minutes After Start
Description: For participants in the experimental (virtual reality) arm, whether the patient completed 20 minutes of use of the ReCognition VR-based software
Time Frame: 20 minutes after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
Participants | 15

14. Other Pre Specified Outcome: Number of Participants With a System Usability Scale (SUS) Score >35
Description: For participants in the experimental (virtual reality) arm, the number of participants with a System Usability Scale (SUS) score >35 on a scale of 0-100, where 0 is minimum and 100 is maximum; higher scores mean better usability.
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
Participants | 12

15. Other Pre Specified Outcome: Proportion of Participants Completing Game With No Errors
Description: The proportion of participants in the experimental (virtual reality) arm who complete the virtual reality game without any user errors
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
Participants | 3

16. Other Pre Specified Outcome: Number of Participants Completing Game on First Attempt
Description: For participants in the experimental (virtual reality) arm, the number of participants who complete the virtual reality game in easy mode on the first attempt
Time Frame: After completion of use of the virtual reality software, up to 2 hours after the start of software use
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software
Number analyzed (Participants) | 15
Participants | 15

17. Post Hoc Outcome: Change in Virtual Analog Scale (VAS) Pain Score From Pre-virtual Reality Use to 10 Minutes After Beginning Use (Experimental Arm) or Enrollment to 8-16 Hours Post-enrollment (Control Arm)
Description: Whether change in VAS pain score using numeric pain rating scale, where 0 is minimum (no pain) and 10 is maximum (highest pain), from pre-virtual reality use to mid-intervention (experimental)/observation (control), grouped by whether the pain score increased, stayed the same (no change), or decreased
Time Frame: Virtual Reality Software arm: 10 minutes after beginning use; Traditional Orientation Methods arm: at 8-16 hours after enrollment (one measure, window allowed for completing the measure)
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
Number analyzed (Participants) | 15 | 15
Participants
  Reduced | 4 | 2
  No Change | 11 | 6
  Increased | 0 | 7
Statistical Analysis 1: Comparison: Virtual Reality Software vs Traditional Orientation Methods; Test type: Superiority; p = 0.011, Fisher Exact

ADVERSE EVENTS:
Time Frame: From the time of surgery to the time the patient was discharged from the hospital, up to 3 months after hospital admission
Arm/Group | Virtual Reality Software | Traditional Orientation Methods
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT06232317/Prot_SAP_000.pdf